CLINICAL TRIAL: NCT03517163
Title: The Boston Outcomes of Autism in Toddlers Study
Brief Title: Boston Outcomes of Autism in Toddlers Study
Acronym: BOAT
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Harstad, Pediatrician, Boston Children's Hospital
Other Study IDs: P00026909
Record Dates: First submitted 2018-04-13; First posted 2018-05-07 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Asperger's; autism; autism spectrum disorder; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Group: Individuals enrolled or just finished kindergarten who were diagnosed with Autism Spectrum Disorder through the DSM-5 diagnostic criteria

SUMMARY:
The purpose of this research study is to learn more about the outcomes of children who received an Autism Spectrum Disorder (ASD) diagnosis when they were toddlers. The study is interested in whether an early diagnosis can help children with their cognitive, language, social, and behavioral abilities.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by deficits in domains of social communication and restrictive and repetitive behavior. There is general agreement, in light of knowledge around optimal periods of neural plasticity, that ASD should be diagnosed as early as possible since young toddlers are at a critical stage in early development when intervention is theoretically most effective. The rate of persistence of an ASD diagnosis is heavily debated.Therefore this study attempts:

1. To determine the rate of persistence of Autism Spectrum Disorder (ASD) diagnosis and functional outcomes, as defined by cognitive level, adaptive functioning, language skills, persistence of ASD symptoms, and classroom placement at kindergarten age, among children who received a DSM-5 ASD diagnosis at < 36 months.
2. To evaluate predictors of rate of persistence and functional outcomes among kindergarten grade level children ages 5-7 years, who received an ASD diagnosis as toddlers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Autism Spectrum Disorder as a toddler through DSM-5 at Boston Children's Hospital
* Enrolled in or just finished Kindergarten

Exclusion Criteria:

* Individuals with known genetic disorders including, but not limited to, Fragile X syndrome, Down syndrome, Tuberous Sclerosis Complex and those with 16 p deletions/duplications.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with Autism Spectrum Disorder through the DSMV as toddlers.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
ASD Symptomatology | 3 years (Age of diagnosis to Kindergarten Age)
  The severity of ASD symptoms in the child (Autism Diagnostic Observation Schedule and Autism Diagnostic Interview-Revised)
Cognitive Level | 3 years (Age of diagnosis to Kindergarten Age)
  Play-based assessment in which a child's cognitive level is determined. (Differential Ability Scales - Second Edition)
Language Level | 3 years (Age of diagnosis to Kindergarten Age)
  Play-based assessment in which a child's language level is determined.Preschool Language Scale - Fifth Edition
Adaptive Functioning | 3 years (Age of diagnosis to Kindergarten Age)
  Parent report on the child's current adaptive functioning (Vineland Adaptive Behavior Scales-3)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Harstad, MD, MPH, Principal Investigator — Pediatrician/Researcher
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States